Assessing the Impact of Herbal Supplement on Fatigue and Disease Activity in SLE: **Results from an 8-Week Randomized Trial** 20-01-2026

### Introduction

Systemic lupus erythematosus (SLE) is a chronic auto-immune disease with a wide range of clinical manifestations and a complex pathogenesis. Despite advancements in treatments for disease activity, fatigue continues to be one of the most prominent and unresolved complaints among patients [1].

According to Jianhua Shen et al. [2], fatigue is defined as an overwhelming sense of tiredness, a lack of energy, and a feeling of exhaustion that is associated with impaired physical and/or cognitive functioning. The prevalence of fatigue in SLE may reach up to 90%, according to some studies[3]. Moreover, over 50% of patients report it as their most disabling symptom[3]. Stress, depression, pain, disease activity, and disease duration are among the most common contributors to fatigue in these patients. Fatigue significantly impacts quality of life (QoL) across all domains physical, psychological, and socio-occupational. Management recommendations for fatigue typically involve a combination of pharmacologic and nonpharmacologic approaches; however, no specific medications have been shown to be effective in treating fatigue associated with SLE[4].Hence, it is essential to evaluate and identify potential intervention areas to alleviate patients' symptom burden and enhance their overall quality of life.

Therefore, we opted for the dietary supplement EVACUR.It is a dietary supplement designed to help combat fatigue and boost the immune system. It combines natural extracts, vitamins, and selenium to support overall vitality.

The aim of our double-blind, placebo-controlled randomized trial was to evaluate the efficacy of using herbal-based treatment on patients with SLE-related fatigue.

### **Methods:**

# **Study Type:**

This was a randomized, double-blind clinical trial conducted in two internal medicine departments in Tunisia over a period of 3 months.

### **Study Population:**

Patients with a diagnosis of SLE who were being followed in the participating departments.

### Inclusion Criteria:

- Age > 18 years
- Confirmed diagnosis of SLE according to the 2019 ACR/EULAR classification criteria
- Presence of fatigue, defined as a FACIT-F score < 34
- Signed informed consent

### Non-Inclusion Criteria:

- Pregnancy or breastfeeding
- Diseases or comorbidities that may influence fatigue:untreated hypothyroidism, psychosis
   common infections, and other autoimmune and inflammatory diseases
- Patients on vitamin K antagonist therapy, due to a possible interaction with Ginger and Nigella
- History of severe allergy or intolerance to EVACUR or any component of the placebo

### Exclusion Criteria:

- Diagnosis of another systemic disease during the study period
- Pregnancy
- Allergy to any component of EVACUR
- Withdrawal of consent

### **Data Collection:**

Patient data were collected from medical records, including epidemiological characteristics such as age at inclusion, gender and medical and family history. Disease-specific data included the duration disease,

systemic manifestations, nature of treatement at inclusion . Disease activity was evaluated using clinical

SLEDAI-2K score. Baseline FACIT score was collected. Biological assessments were performed such

us Anti-dsDNA antibody titers ,ANA and serum C3 and C4 levels.

**Study protocol:** 

**Randomization:** 

A two -to-one (2:1) randomization was performed in this study in which patients were randomly

assigned into two groups: Group 1 (G1) which received EVACUR, and Group 2 (G2) received a

placebo. Randomization was handled by an independent third party using a dedicated randomization

software.

**Double-Blind Design:** 

Neither the patients nor the investigators knew the treatment assignment. EVACUR and placebo

capsules are identical in appearance.

**Treatement:** 

**EVACUR**:

A phytotherapeutic compound presented in capsule form. Each bottle contains 40 capsules composed

of: Nigella seed, Zinc sulfate, Echinacea, Vitamin C, Red ginseng, Ginger, Chamomile, Spirulina, Royal

jelly, Ganoderma, Vitamins B1, B6, B12, Selenium(Table1).

Contra-indications: Allergy to any component of the supplement.

Placebo:

Capsules containing starch, packaged identically to EVACUR bottles.

Both treatments will be administered at a dose of 2 capsules per day in the morning (3 bottles per

patient for the study duration).

Follow-up:

Patients attended three visits at baseline M0, one month M1, and two months M2. The FACIT score

was assessed during each visit along with a physical examination.

**Adverse Events:** 

Potential side effects will be recorded and evaluated throughout the study. Occurrence of any adverse

event will lead to patient exclusion and trigger a pharmacovigilance investigation. All adverse events

must be reported immediately to the principal investigator.

**Fatigue Assessment Score:** 

Functional Assessment of Chronic Illness Therapy – Fatigue (FACIT-F)

A 13-item questionnaire with responses on a Likert scale from 1 (not at all) to 5 (very much).

Total score out of 52; higher scores indicate less fatigue. Can be calculated if at least 50% of the

questions are answered.

**Reliability**: High (Cronbach's alpha = 0.94)

Validity: Strong, with good correlation with other fatigue measurement tools

Completion time: 5–10 minutes

A validated Arabic version is available with good psychometric properties .

**Evaluation Criteria:** 

**Primary Endpoint:** 

A mean Facit-F score improvement between G1 and G2 at month2 > Minimal Clinically Important

Difference(MCID). The MCID in SLE is estimated at 3.4T[5].

## **Secondary Endpoints:**

Improvement in the disease activity SLEDAI score

Good tolerance of the dietary supplement.

### **Statistical Analysis:**

Data were analyzed using SPSS.Appropriate statistical tests will be applied, including Student's t-test or the Wilcoxon test.Randomization will be conducted using dedicated software.

#### **Ethical considerations**

This study was conducted according to the Declaration of Helsinki and approved as well by the RABTA hospital's ethics committee under the number of CERB33/2023. Informed consent was given by each patient before starting the study. Each patient will be assigned an inclusion number used for randomization and data entry, ensuring patient confidentiality.

## **Statements & declarations:**

- **Funding**: Wellnet Pharmaceutical Factory ® provided the dietary supplement and the placebo free of charge.No additional funding was required
- Conflict of Interest: Wellnet Pharmaceutical Factory® had no role in the study design, data collection, analysis, interpretation, or decision to submit the manuscript for publication.

### -Informed consent

Informed consent was obtained from all individual participants included in the study after reading and agreeing with the details of this trial.

- Availability of data and material :data are available on request from the authors
- **Ethics approval**: Patients' anonymity was maintained throughout the study. The study was approved by the ethics committee of the hospital under the number CERB 33/2023.

 Table 1. Ingredients and Dosage of EVACUR Formulation per Capsule

| Ingredient | Latin/INCI Name | Form/Quality | Quantity per capsule |
|---|---|---|---|
| Black seed | Nigella sativa | Dry extract | 80 mg |
| Echinacea | Echinacea spp. | Dry extract | 40 mg |
| Ginger | Zingiber officinale | Dry extract | 30 mg |
| Chamomile | Matricaria chamomilla | Dry extract | 10 mg |
| Red ginseng | Panax ginseng | Dry extract | 10 mg |
| Reishi mushroom | Ganoderma lucidum | Dry extract | 10 mg |
| Spirulina | Spirulina spp. | Dry extract | 60 mg |
| Royal jelly | Royal jelly | Lyophilized | 20 mg |
| Vitamin C | Ascorbic acid | | 30 mg |
| Zinc | Zinc sulfate | | 2.5 mg |
| Vitamin B1 | Thiamine | _ | 3 mg |
| Vitamin B6 | Pyridoxine | Marine source | 4 mg |
| Vitamin B12 | Cobalamin | | 10 μg |
| Selenium | Selenium yeast | _ | 40 μg |